CLINICAL TRIAL: NCT07309172
Title: Keto-Brain: Cerebral Energy Substrate Metabolism in First-Episode Schizophrenia
Brief Title: KetoBrain: Brain Energy Metabolism in Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: Ole Köhler-Forsberg (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ole Köhler-Forsberg, MD, PhD, Assoc. Professor, University of Aarhus
Organization: University of Aarhus (Other)
Other Study IDs: 2025_KetoBrain
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia Disorder
Keywords: Schizophrenia; PET neuroimaging; Brain energy substrate metabolism; Ketone bodies; Glucose
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be stored at -80 C to measure ketone bodies. After this, the blood samples will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with first-episode schizophrenia
- Healthy controls

SUMMARY:
Objective The objective is to recruit antipsychotic-naïve patients at the first diagnosis with a first-episode schizophrenia disorder (FES) to study ketone metabolism of the brain via PET neuroimaging. Participants will undergo PET neuroimaging at baseline before start of antipsychotic treatment and after 4-8 weeks of antipsychotic treatment including an additional clinical follow-up visit after 6 months. In addition, a healthy control group with one baseline visit will be recruited.

Study design Non-interventional neuroimaging study with pre-defined follow-up visits.

Patients Patients with a FES (ICD-10: F20) aged 18-35 years who are antipsychotic-naïve including age- and sex-matched healthy controls.

Sample size This is an observational pilot project. Currently, no studies have measured brain ketone metabolism before and after AP intake. Assuming a 50% dropout rate at follow-up, the investigators aim to recruit 22 patients to obtain 12 full datasets - a sample size commonly used in PET studies. Healthy controls will only have one study day, so no dropouts are expected - aiming at a sample size of 12 healthy controls.

Procedures Patients will be included at the first FES diagnosis. Before inclusion, an interview with the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview will validate the diagnosis. At baseline and follow-up (details in the full protocol and Table 1), patients will be rated by use of the 6-item Positive and Negative Syndrome Scale (PANSS-6), the Clinical Global Impression Severity Scale (CGI-S), the Global Assessment of Functioning Scale (GAF), Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT), Fagerström Test for Nicotine Dependence (FTND), and the Calgary Depression Scale for Schizophrenia (CDSS). The Matrics Consensus Cognitive Battery (MCCB), which consists of 10 cognitive tests, will measure cognition. Heart rate, blood pressure, height, body weight, waist and hip circumference will be recorded. Patients will be treated according to clinical indication, i.e., they will receive routine clinical care at the local psychiatric hospital and participation in this study will not affect the treatment.

Follow-up Patients will be treated and followed according to normal clinical treatment guidelines at the local psychiatric hospitals, which will not be affected by participation. A re-scan will be performed after 4-8 weeks of antipsychotic treatment.

Endpoints The primary endpoints are

1. Brain ketone and glucose metabolism in FES before antipsychotic treatment compared to healthy controls measured via PET
2. Brain ketone and glucose metabolism in FES after antipsychotic treatment

Risks and Safety Patients will follow treatment-as-usual at their local psychiatric hospital, with the clinicians from the local hospital being responsible for safety monitoring according to local treatment guidelines. Participation in the present study will not delay clinically indicated antipsychotic treatment. Blood sample results will be obtained from the patient's medical record (MidtEPJ) at the study visits to monitor biochemical safety parameters for medical treatment. Between follow-up visits for this study, patients will follow guideline-based safety monitoring at the local psychiatric hospital.

During the PET neuroimaging, participants will have two catheters, one arterial and one venous. Vascular puncture can result in a light degree of pain. The risk of infection is negligible.

PET: Injection of the radiotracer may cause slight pain and redness, which should rapidly resolve. The radiotracers [15O]H2O and [11C]OHB are radiolabeled versions of their naturally occurring versions, thus sharing their chemical properties. They are given in non-pharmacological doses. [18F]FDG is an analogue of glucose, given in non-pharmacological dose (<1 nanogram). Allergic reactions have been described, but are extremely rare - it has been used routinely in the workup of cancer patients through decades. Ultimately, no pharmacologic or immunologic side effects are to be expected from the radiotracers.

The amount of radiation to healthy controls will be 4.6 mSv. Since patients have two study days, the total radiation dose to patients will be 9.2 mSv. The mean background radiation in Denmark is approximately 3 mSv per year. Thus, healthy subjects and patients will get approximately 1½ and 3 times the yearly background radiation during the study. In Denmark, the lifetime risk of lethal cancer is approximately 25%. The radioactive dose of 9.2 mSv administered to patients in this study, may increase the risk by 0.05% (from 25% to 25.05%). The radioactive dose of 4.6 mSv administered to healthy controls in this study, may increase the risk by 0.02% (from 25% to 25.02%).

Study duration 2025-2027.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with FES

1. Age 18-35 years
2. Diagnosed with FES (ICD-10: F20)
3. Able to give informed oral and written consent.

Inclusion criteria for healthy controls

1. Age 18-35 years
2. No mental disorder (ICD-10: F00-99)
3. Able to give informed oral and written consent.

Exclusion Criteria:

Exclusion criteria for patients with FES

1. Any coercive measure including patients in forensic psychiatry
2. In a clinical condition where the treating clinician evaluates that the patient is not able to attend the research study.
3. Previous use of AP at an antipsychotic dose (except for Risperidone ≤0.5 mg, Abilify ≤2.5 mg, Seroquel ≤50 mg or Zyprexa ≤2.5 mg) for more than 2 continuous weeks in the past year and/or 6 weeks over a lifetime
4. Use of an antipsychotic in the last 3 months before inclusion at a dose greater than:

   4.1 Seroquel/Quetiapine 50 mg 4.2 Risperdal/Risperidone 0.5 mg
5. Comorbidity: Borderline intelligence or intellectual disability, autism spectrum disorder, decompensated substance use disorder, psychosis induced by a medical condition or psychosis induced by medication or drug use.
6. Pregnancy, childbirth within the past 6 months, or breastfeeding. Female participants should use an effective contraception.
7. Contraindications to MRI (metal, severe claustrophobia).
8. Acute suicidal thoughts (e.g., resulting in hospitalization)
9. Diabetes mellitus type 1. History of severe head trauma, stroke, chemotherapy or brain surgery. Hypo- or hyperthyroidism. Epilepsy. Systemic glucocorticoid hormone treatment.
10. Other conditions interfering with participation according to the qualified physician's judgment.

Exclusion criteria for healthy controls

1. Previous use of an antipsychotic dose (except for Risperidone ≤0.5 mg, Abilify ≤2.5 mg, Seroquel ≤50 mg or Zyprexa ≤2.5 mg) for more than 2 continuous weeks in the past year and/or 6 weeks over a lifetime
2. Use of AP in the last 3 months before inclusion at a dose greater than:

   1. Seroquel/Quetiapine 50 mg
   2. Risperdal/Risperidone 0.5 mg
3. Pregnancy, childbirth within the past 6 months, or breastfeeding. Female participants should use an effective contraception.
4. Contraindications to MRI (metal, severe claustrophobia).
5. Diabetes mellitus type 1. History of severe head trauma, stroke, chemotherapy or brain surgery. Hypo- or hyperthyroidism. Epilepsy. Systemic glucocorticoid hormone treatment.
6. Other conditions interfering with participation according to the qualified physician's judgment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Antipsychotic-naive patients with FES and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole brain ketone and glucose metabolism in FES compared to healthy controls measured via PET | At enrollment, i.e. at the baseline PET scan
Whole brain ketone and glucose metabolism in FES after antipsychotic treatment | From baseline scan to the follow-up scan after 4-8 weeks of antipsychotic treatment

SECONDARY OUTCOMES:
Correlation between antipsychotic response, as measured on the PANSS-6, with the change in brain ketone and glucose metabolism in patients with FES | From baseline to follow-up scan after 4-8 weeks of antipsychotic treatment
Correlation between the MCCB with the change in brain ketone and glucose metabolism in patients with FES | From baseline to follow-up scan after 4-8 weeks of antipsychotic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Psychosis Research Unit, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No